CLINICAL TRIAL: NCT00550459
Title: A Pilot, Phase 3B, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study of the Effects of Titrated Oral Tolvaptan 15, 30, or 60 mg QD on Cognitive and Neurological Function in Elderly Hyponatremic Patients
Brief Title: Effects of Titrated Oral Tolvaptan 15-60 mg Once Daily (QD) on Cognitive and Neurological Function in Elderly Hyponatremic Patients
Acronym: INSIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Dorothee Oberdhan, Manager, Global Clinical Development, Otsuka Pharmaceutical Development & Commercialization, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-04-246; INSIGHT
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Results first posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Cognitive; Neurological Function; Elderly
MeSH Terms: conditions — Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo tablet given once a day for 21 days
  Interventions: Drug: Placebo
- 2 (Active Comparator): Tolvaptan 15 mg-60 mg tablet given once a day for 21 days.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — 15-60 mg oral tablet given once a day for 21 days.
  Other Names: OPC-41061
  Arms: 2
Drug: Placebo — Placebo tablet given once daily for 21 days
  Arms: 1

SUMMARY:
Demonstrate an improvement in the composite scores of validated neurocognitive tests in elderly subjects with chronic sub-clinical (i.e., asymptomatic) hyponatremia.

DETAILED DESCRIPTION:
Subjects will be randomized, with stratification by baseline sodium <130 or ≥ 130 mEq/L[mmol/L] to receive either tolvaptan 15 mg tablet or matching placebo tablet at doses of 15, 30 or 60 mg for 21 days. During this period, fluid restrictions should be loosened or suspended, until the subject's response to therapy can be evaluated, typically over the first few days of therapy. Fluid restriction may be reinstituted at any time in subjects whose sodium fails to improve or worsens with study therapy. A forced-titration up to 60 mg of study drug by day 3 to 7 will be based on the subject's serum sodium Subjects entering the study with a serum sodium concentration less than 130 mEq/L[mmol/L] may be fluid restricted if necessary at the discretion of the Investigator. Subjects should be monitored closely during the first 24 hours of treatment for dosing titration. The total dosing duration will be up to 21 days (plus 3 day treatment window). Subjects will return to the clinic on Day 22 (+3 days) for assessments and will complete a follow-up visit on Day 28 (+2 days).

ELIGIBILITY:
Inclusion Criteria:

* Women and men 50 years of age or older.
* Serum Sodium ≥123 and ≤ 134 mEq/L [mmol/L]at screening and baseline.
* Subjects with serum sodium concentrations ≥118 and ≤122 mEq/L[mmol/L] at screening and baseline may be entered into the trial based on consultation and approval from the study medical monitor.

Exclusion Criteria:

* Conditions or history which may present a safety concern to the subject or their offspring or extreme susceptibility to hypotension with sudden fluid loss (aquaresis).
* Hyponatremia that is acute, easily reversible, artifactual, or due to a condition not associated with vasopressin excess or likely to respond to aquaretic therapy.
* Conditions associated with an independent imminent risk of morbidity and mortality.
* Conditions which may confound the assessment of endpoints, history of poor compliance, participation in a clinical trial believed by the PI or Sponsor likely to confound endpoint assessments.
* Conditions which may confound primary endpoints of cognitive function.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Verbalis, MD, Principal Investigator — Georgetown University, Washington, DC, 20007 USA
Locations (12):
- United States (12):
  - Sarah. S. Olelewe, MD, Hawthorne, California
  - Progressive Clinical Research, Vista, California
  - Pikes Peak Cardiology, Colorado Springs, Colorado
  - Innovative Research of West FL, Largo, Florida
  - Coastal Nephrology Assoc. Research Center, Punta Gorda, Florida
  - Rockdale Medical Research Associates, Conyers, Georgia
  - Otis Barnum, DO, Natchitoches, Louisiana
  - Lillestol Research, LLC, Fargo, North Dakota
  - Carolina Research Associates, Columbia, South Carolina
  - Wayne O. Wells, MD, Lebanon, Tennessee
  - Memorial Clinical Associates, Houston, Texas
  - Mitchell Rosner, MD, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 United States (US) sites/clinics; first subject signed informed consent on 9/11/07; last subject's final visit on 12/16/08
Groups:
- Tolvaptan (15-60 mg): Tolvaptan tablet 15-60 mg given once daily for 21 days
Period: Overall Study
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Started | 28 | 29
Completed | 27 | 26
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tolvaptan (15-60 mg) | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 22 | 23 | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 71.3 (9.7) | 71.1 (10.2) | 71.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 9 | 14 | 23
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Neurocognitive Composite Score of Speed Domains (NCS-SD; Sum of All Correct Speed Domain Z-Scores)
Description: Change from baseline to Day 22 in sum of all speed domain Z-scores:Reaction Time (Simple=recognize "yes" 50 times;Choice=recognize "yes" or "no" 50 times;Digit Vigilance=match 45 digits);Psychomotor Speed (Morse Tapping=tap button for 30 seconds with right & left hands);Processing Speed (Rapid Visual Information Processing=detect consecutive sequences of 3 odd or 3 even digits;Numeric Working Memory=recognize numbers from series of 5 digits among 30;Word Recognition=remember 15 prior learned words from 30 total;results age-matched to healthy controls from Cognitive Drug Research normative data
Time Frame: baseline and Day 22
Population: Analysis based upon observed cases (OC).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 27 | 26
Z-score | 0.20 (0.61) | 0.39 (0.49)
Statistical Analysis 1: Comparison: Placebo vs Tolvaptan (15-60 mg); Analysis of covariance (ANCOVA) with factors of treatment,disease severity (<130mEq/L [mmol/L] or ≥130mEq/L [mmol/L] at baseline),age (<65, ≥65 to <75,and ≥75 years) (factor with 6 Degrees of Freedom), and covariate baseline used to fit primary endpoint using the intent-to-treat (ITT) dataset. Estimated treatment effect and its 95% confidence interval (CI) provided under the model with p-value. A 2-sided alpha (0.05) applied to the primary analysis. Primary analysis based on observed cases (OC); Test type: Superiority or Other; p = 0.08, ANCOVA — Secondary endpoints were ordered in 5 tiers to be analyzed only when >=1 of the endpoints in the prior tier were significant. Since primary endpoint not stat significant, analyses of secondary endpoint tiers presented for exploratory purposes only; ANCOVA with factors of treatment, disease severity, age(6 Degrees of Freedom), and covariate baseline to fit primary endpoint using the ITT dataset; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.03 to 0.50], Standard Deviation 0.55

2. Secondary Outcome: Change From Baseline to Day 22 in the Individual Neurocognitive Domains Included in the Primary Endpoint: Reaction Time in Computer Tests
Description: Change from baseline in the individual neurocognitive domains Z-score for Reaction Time in Computer Tests (simple reaction time test, choice reaction time test, digit vigilance test); ITT population
Time Frame: baseline and Day 22
Population: ITT population with OC
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 27 | 26
Z-score | 0.21 (0.86) | 0.33 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Tolvaptan (15-60 mg); Per-protocol, secondary endpoints were ordered in 5 tiers and were to be analyzed only when at least 1 of the endpoints in the previous tier was significant. As the primary endpoint was not statistically significant, the analyses of subsequent secondary endpoint tiers are presented for exploratory purposes only; Test type: Superiority or Other; p = 0.21, ANCOVA — ANCOVA with factors of treatment, disease severity, age, and severity by age interaction, and baseline as covariate. The estimated treatment and its 95% CI were provided under the model along with the p-value; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.12 to 0.51], Standard Deviation 0.63

3. Secondary Outcome: Change From Baseline in the Individual Neurocognitive Domains Included in the Primary Endpoint: Psychomotor Speed Via Morse Tapping Test
Description: Change from baseline to Day 22 in the individual neurocognitive domains Z-score for Psychomotor Speed (mean tap rate of Morse tapping test); ITT population
Time Frame: baseline and Day 22
Population: ITT population with OC
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 27 | 26
Z-score | 0.04 (0.36) | 0.31 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Tolvaptan (15-60 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.02, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Median Difference (Net) = 0.27, 95% CI 2-sided [0.04 to 0.51], Standard Deviation 0.41

4. Secondary Outcome: Change From Baseline in the Individual Neurocognitive Domains Included in the Primary Endpoint: Processing Speed of Rapid Visual Information Processing Test, Numeric Working Memory Test, and Word Recognition Test
Description: Change from baseline to Day 22 in the individual neurocognitive domains Z-score for Processing Speed of Rapid Visual Information Processing Test, Numeric Working Memory Test, and Word Recognition Test; ITT population
Time Frame: baseline and Day 22
Population: ITT population with OC
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 27 | 26
Z-score | 0.24 (0.75) | 0.48 (0.91)
Statistical Analysis 1: Comparison: Placebo vs Tolvaptan (15-60 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.21, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.15 to 0.67], Standard Deviation 0.83

5. Secondary Outcome: Change From Baseline in Overall Neurocognitive Composite Score
Description: Change from Baseline to Day 22 in the overall Neurocognitive Composite Score (NCS)comprising the sum of 7 neurocognitive domain Z-scores (Reaction Time, Psychomotor Speed, Processing Speed, Continuity of Attention, Working Memory/Executive Functions, Quality of Episodic Verbal Memory, and Postural Stability); ITT population
Time Frame: baseline and Day 22
Population: ITT population with OC
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 27 | 26
Z-score | 0.19 (0.39) | 0.30 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Tolvaptan (15-60 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.16, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.05 to 0.30], Standard Deviation 0.39

6. Secondary Outcome: Change From Baseline in Gait Test (Timed Get-Up-and-Go Test)
Description: Change from baseline to Day 22 in Gait Test (Timed Get-Up-and-Go Test=time it takes for a seated subject to rise from a chair, walk 3 meters, walk around an object and return to sit in chair. Values: under 10 sec (no difficulties), 10 to 20 sec (starting to have balance difficulty), over 30 sec (at high risk for falls and dependent in most activities of daily living and mobility); test assesses risk to elderly subjects of falling and higher scores in seconds indicate higher risk of falling; ITT population
Time Frame: baseline and Day 22
Population: ITT population with OC
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 26 | 23
Seconds | 1.06 (5.63) | -0.43 (1.54)
Statistical Analysis 1: Comparison: Placebo vs Tolvaptan (15-60 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.23, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = -1.51, 95% CI 2-sided [-4.02 to 1.00], Standard Deviation 3.53

7. Secondary Outcome: Change From Baseline in Postural Stability Test
Description: Change from baseline to Day 22 in Postural Stability Test Z-score (This test measures gross motor control. The ability to stand upright without moving is assessed using the SWAY meter that is modeled on the Wright Ataxiameter. A cord from the meter is attached to the subject who is required to stand as still as possible with feet apart and eyes closed for 1 minute. The test is then repeated with eyes open for 1 minute. The outcomes of these tests are combined and measured as a movement Z-score. Higher result=better postural stability); ITT population
Time Frame: baseline and Day 22
Population: ITT population with LOCF (this group includes missing values)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 25 | 23
Z-score | 1.3 (4.68) | -0.35 (2.33)
Statistical Analysis 1: Comparison: Placebo vs Tolvaptan (15-60 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.18, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.83, 95% CI 2-sided [-2.04 to 0.38], Standard Deviation 3.51

8. Secondary Outcome: Change From Baseline in Serum Sodium; ITT Population
Description: Change from Baseline to Day 22 in Serum Sodium; ITT population
Time Frame: Baseline and Day 22
Population: ITT population with OC
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 26 | 26
mEq/L | 2.23 (3.51) | 7.04 (3.39)
Statistical Analysis 1: Comparison: Placebo vs Tolvaptan (15-60 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 4.75, 95% CI 2-sided [2.89 to 6.60], Standard Deviation 3.45

9. Secondary Outcome: Number of Patients With Vital Sign Abnormalities: Blood Pressure
Description: Incidence of abnormal systolic & diastolic blood pressure values post-baseline (abnormal systolic values: >=180 mmHg + increase of >=20 mmHg, <= 90 mmHg + decrease >=20 mmHg; abnormal diastolic values: >=105 mmHg+increase of >=15 mmHg, <=50 mmHg + decrease of >= 15 mmHg)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 2 | 0

10. Secondary Outcome: Number of Patients With Vital Sign Abnormalities: Pulse Rate
Description: Incidence of abnormal pulse rate post-baseline [abnormal values: >=120 beats per minute (bpm) + increase of >=15 bpm; <=50 bpm + decrease of >=15 bpm]
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 0 | 0

11. Secondary Outcome: Number of Patients With Vital Sign Abnormalities: Body Weight
Description: Incidence of clinically significant body weight change post-baseline (defined as change upward or downward of >=7%)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 27 | 29
participants | 1 | 1

12. Secondary Outcome: Number of Patients With Vital Sign Abnormalities: Body Temperature
Description: Incidence of potentially clinically significant changes in body temperature post-baseline (defined as an increase of >=1.1 to >=38.3 degrees Celsius)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 1 | 0

13. Secondary Outcome: Number of Patients With Hematology Laboratory Abnormalities: Hemoglobin
Description: Incidence of clinically significant hemoglobin abnormalities post-baseline (normal range=11.8-16.8 g/dL)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 26 | 29
participants | 0 | 1

14. Secondary Outcome: Number of Patients With Hematology Laboratory Abnormalities: Activated Partial Thromboplastin Time (aPTT)
Description: Incidence of potentially clinically significant Activated Partial Thromboplastin Time (aPTT) levels post-baseline (normal range=22-34 seconds)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 27 | 29
participants | 1 | 3

15. Secondary Outcome: Number of Patients With Hematology Laboratory Abnormalities: Lymphocytes
Description: Incidence of potentially clinically significant lymphocyte count post-baseline (normal range = 16-46%)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 26 | 29
participants | 1 | 2

16. Secondary Outcome: Number of Patients With Hematology Laboratory Abnormalities: Neutrophils
Description: Incidence of potentially clinically significant neutrophil count post-baseline (normal range=1.8-8 thousands/microliter)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 26 | 29
participants | 2 | 0

17. Secondary Outcome: Number of Patients With Serum Chemistry Laboratory Abnormalities: Blood Urea Nitrogen (BUN)
Description: Incidence of potentially clinically significant BUN levels post-baseline (normal range=7-30 mg/dL)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 1 | 2

18. Secondary Outcome: Number of Patients With Serum Chemistry Laboratory Abnormalities: Uric Acid
Description: Incidence of potentially clinically significant uric acid levels post-baseline (normal range=4-8.5 mg/dL)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 0 | 1

19. Secondary Outcome: Number of Patients With Serum Chemistry Laboratory Abnormalities: Cholesterol
Description: Incidence of potentially clinically significant cholesterol levels post-baseline (normal range=0-199 mg/dL)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 0 | 2

20. Secondary Outcome: Number of Patients With Serum Chemistry Laboratory Abnormalities: Glucose
Description: Incidence of potentially clinically significant glucose levels post-baseline (normal range=70-125 mg/dL)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 2 | 0

21. Secondary Outcome: Number of Patients With Serum Chemistry Laboratory Abnormalities: Magnesium
Description: Incidence of potentially clinically significant magnesium levels post-baseline (normal range=1.2-2 mEq/L)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 0 | 1

22. Secondary Outcome: Number of Patients With Electrocardiogram (ECG) Abnormalities: QT >500 Milliseconds (Msec)
Description: Incidence of potentially clinically significant ECG abnormalities (QT>500 msec) post-baseline
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 1 | 0

23. Secondary Outcome: Number of Patients With Electrocardiogram (ECG) Abnormalities: QRS Interval
Description: Incidence of potentially clinically significant ECG abnormalities involving QRS interval (change > 100 msec)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 1 | 1

24. Secondary Outcome: Number of Patients With Electrocardiogram (ECG) Abnormalities: QTcB Increase 30-60 Msec
Description: Incidence of potentially clinically significant ECG abnormalities (QTcB increase 30-60 msec)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 3 | 4

25. Secondary Outcome: Number of Patients With Electrocardiogram (ECG) Abnormalities: QTcF Increase 30-60 Msec
Description: Incidence of potentially clinically significant ECG abnormalities (QTcF increase 30-60 msec post-baseline)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 2 | 3

26. Secondary Outcome: Number of Patients With Electrocardiogram (ECG) Abnormalities: ST Segment
Description: Incidence of potentially clinically significant ECG abnormalities: ST Segment
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 0 | 2

27. Secondary Outcome: Number of Patients With Electrocardiogram (ECG) Abnormalities: T Wave
Description: Incidence of potentially clinically significant ECG abnormalities: T wave
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 1 | 1

28. Secondary Outcome: Number of Patients With Electrocardiogram (ECG) Abnormalities: Right Bundle Branch Block (RBBB), Left Bundle Branch Block (LBBB), Myocardial Infarction (MI)
Description: Incidence of potentially clinically significant ECG abnormalities: Right bundle branch block (RBBB), Left bundle branch block (LBBB), myocardial infarction (MI)
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 0 | 1

29. Secondary Outcome: Number of Patients With Electrocardiogram (ECG) Abnormalities: Arrhythmia
Description: Incidence of potentially clinically significant ECG abnormalities: arrhythmia
Time Frame: 28 days
Population: Safety population defined as all randomized subjects who consumed at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Number analyzed (Participants) | 28 | 29
participants | 2 | 6

ADVERSE EVENTS:
Time Frame: 28 Days
Description: collection/elicitation of adverse event incidence
Arm/Group | Placebo | Tolvaptan (15-60 mg)
Serious Adverse Events (participants affected / at risk) | 1/28 | 2/29
Other Adverse Events (participants affected / at risk) | 13/28 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Tolvaptan (15-60 mg) (N=29)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Tolvaptan (15-60 mg) (N=29)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 3 (4) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 4 (4)
Thirst (General disorders) | 2 (2) | 6 (6)
Urine output increased (Investigations) | 0 (0) | 3 (3)
Weight decreased (Investigations) | 0 (0) | 4 (4)

LIMITATIONS AND CAVEATS:
Pilot study powered only for serum Na+ improvements. Trial lacked sufficient power to detect changes in neurocognitive test scores and SF-12 and HDS outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No